CLINICAL TRIAL: NCT07086417
Title: A Prospective Controlled Study on Robot-Assisted Versus Conventional Arthroscopic Anterior Cruciate Ligament Reconstruction
Brief Title: Robot-Assisted Versus Conventional Arthroscopic ACL Reconstruction: A Prospective Comparative Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chunyan Jiang (Other)
Collaborators: Star Sports Medicine Co., Ltd (Unknown)
Responsible Party: Sponsor-Investigator, Chunyan Jiang, Director of the Department of Sports Medicine, Beijing Jishuitan Hospital
Organization: Beijing Jishuitan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Z221100007422004
Record Dates: First submitted 2025-07-18; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Anterior Cruciate Ligament

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robot-Assisted ACL Reconstruction (Experimental): Participants in this group will undergo arthroscopic anterior cruciate ligament (ACL) reconstruction using a custom-designed robotic surgical system. The system includes preoperative planning, intraoperative guidance, and biomechanical evaluation modules. Tunnel positions are planned based on CT and MRI fusion images, and the robot assists the surgeon with precise femoral and tibial tunnel drilling. Biomechanical assessments such as graft isometry and impingement risk are evaluated intraoperatively.
  Interventions: Procedure: Robot-Assisted Arthroscopic ACL Reconstruction
- Conventional Arthroscopic ACL Reconstruction (Active Comparator): Participants in this group will receive conventional arthroscopic ACL reconstruction. Femoral and tibial tunnels are created manually using standard guides and instrumentation. Graft placement and tensioning are performed according to traditional techniques, and isometry and impingement are assessed manually during surgery.
  Interventions: Procedure: Conventional Arthroscopic ACL Reconstruction

INTERVENTIONS:
Procedure: Robot-Assisted Arthroscopic ACL Reconstruction — This intervention involves the use of a customized robotic surgical system to assist in arthroscopic anterior cruciate ligament (ACL) reconstruction. The system integrates preoperative planning with CT/MRI fusion imaging, intraoperative surgical guidance for femoral and tibial tunnel creation, and real-time biomechanical evaluation. The robot provides enhanced precision in tunnel positioning and graft placement compared to conventional techniques.
  Arms: Robot-Assisted ACL Reconstruction
Procedure: Conventional Arthroscopic ACL Reconstruction — This intervention uses standard arthroscopic techniques for ACL reconstruction without robotic assistance. Tunnel positions are determined manually using surgical landmarks and guides. Graft placement, tensioning, and isometry assessment are performed by the surgeon using conventional methods.
  Arms: Conventional Arthroscopic ACL Reconstruction

SUMMARY:
This study aims to evaluate the clinical efficacy and biomechanical accuracy of a newly developed robot-assisted system for anterior cruciate ligament (ACL) reconstruction. ACL injuries are among the most common sports-related injuries in active individuals and athletes, and reconstruction surgery is considered the gold standard for treatment. However, failure rates remain substantial-up to 10.3% in the general population and as high as 40% among high-demand patients, such as young athletes. One of the key technical factors contributing to graft failure is improper placement of the femoral and tibial bone tunnels during surgery, which affects graft isometry, kinematics, and long-term function.

This prospective, randomized, controlled clinical trial will include 120 adult patients with confirmed ACL rupture. Subjects will be randomly assigned to two groups: an experimental group undergoing robot-assisted arthroscopic ACL reconstruction, and a control group receiving traditional arthroscopic ACL reconstruction. The investigational robot system is a custom-designed platform that integrates three primary modules: (1) preoperative planning, (2) intraoperative surgical assistance, and (3) biomechanical evaluation. The robot is designed to support precise tunnel positioning using CT/MRI fusion, dynamic motion tracking during surgery, and post-placement assessment of graft trajectory, potential impingement, and mechanical stability.

Preoperative planning includes 3D reconstruction from CT and MRI imaging to identify optimal anatomical positions for the femoral and tibial tunnels. During surgery, the robot allows the surgeon to perform the procedure in a semi-active "cooperative control" mode, combining robotic precision with the surgeon's decision-making and dexterity. Unlike existing robotic platforms, this system enables limited patient limb movement and real-time position tracking, making it uniquely suited for arthroscopic procedures.

The primary endpoint of the study is anterior tibial translation at 2 years postoperatively, measured using the KT-1000 arthrometer to compare surgical and contralateral knees. Secondary endpoints include subjective knee function scores (Lysholm, Kujala, and Tegner), CT and MRI evaluation of tunnel placement and graft integration, and physical examination results. Follow-up will occur preoperatively and at 2 years postoperatively via in-person visits.

Sample size was calculated based on differences in Lysholm scores from prior navigation-assisted studies. With an alpha level of 0.05, a power of 0.90, and a 20% expected loss to follow-up, 60 patients will be enrolled in each group. Data will be analyzed using SPSS v22.0. Parametric and non-parametric tests will be applied as appropriate, including ANOVA, Bonferroni post-hoc comparisons, and Cochran's Q for repeated categorical variables. A p-value <0.05 will be considered statistically significant.

This study is conducted by the Department of Sports Medicine at Beijing Jishuitan Hospital, a leading orthopedic and trauma care center in China, affiliated with Capital Medical University. The project is supported by the Capital Clinical Special Diagnosis and Treatment Technology Research and Translational Application Program and involves collaboration with Beijing Tiansing Bomed Medical Devices Co., Ltd., which is responsible for the robotic platform development and maintenance.

Ethical approval has been obtained from the Institutional Review Board of Beijing Jishuitan Hospital. All patients will provide written informed consent before enrollment. The study complies with the Declaration of Helsinki, Good Clinical Practice (GCP) guidelines, and local regulations.

Expected outcomes of this study include evidence of improved tunnel placement accuracy, enhanced functional recovery, and potentially reduced failure rates with robot-assisted ACL reconstruction. If successful, this research may contribute to broader adoption of robotic technology in arthroscopic sports medicine surgery and support future innovations in orthopedic surgical robotics.

ELIGIBILITY:
Inclusion Criteria:

* Age over 16 years old; Primary anterior cruciate ligament (ACL) rupture confirmed by physical examination and MRI; Surgery scheduled within 3 months of injury; Patients eligible for autograft ACL reconstruction using 8S-ST/G technique; Normal range of motion in the contralateral knee; Willingness to participate and sign informed consent.

Exclusion Criteria:

* Previous surgery on either knee; Multi-ligament injuries or complex injuries requiring additional procedures; History of rheumatologic or systemic inflammatory joint diseases; Moderate to severe osteoarthritis (Kellgren-Lawrence grade ≥ 2); Poor general health or contraindications to surgery; Refusal to participate or inability to follow up.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Anterior Tibial Translation Measured by KT-1000 | At 24 months post-operation
  Anterior tibial translation will be measured using the KT-1000 arthrometer to assess knee joint stability. The difference in anterior translation between the operated and contralateral knees will be recorded. This outcome is intended to evaluate the functional success of ACL reconstruction and the accuracy of tunnel positioning.

SECONDARY OUTCOMES:
Lysholm Knee Score | Baseline and 24 months post-operation
  Lysholm score will be used to assess knee function and stability. Patients will complete the questionnaire before surgery and at 24 months postoperatively. Scores range from 0 to 100, with higher scores indicating better function.
Kujala Anterior Knee Pain Score | Baseline and 24 months post-operation
  The Kujala score evaluates anterior knee pain and function during activities such as walking, squatting, and climbing stairs. It will be administered preoperatively and 24 months after surgery. Higher scores indicate fewer symptoms.
MRI Evaluation of Graft Position and Integrity | Immediate postoperative period and 24 months post-operation
  MRI will be used to assess the position of the femoral and tibial tunnels and the integrity of the ACL graft. Imaging will be performed immediately after surgery and at 24 months postoperatively.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-03-25): https://cdn.clinicaltrials.gov/large-docs/17/NCT07086417/Prot_SAP_000.pdf
  • Informed Consent Form (2025-03-25): https://cdn.clinicaltrials.gov/large-docs/17/NCT07086417/ICF_001.pdf